CLINICAL TRIAL: NCT06302036
Title: The Effect of Online Emotional Freedom Techniques (EFT) on Stress, Anxiety and Depression in University Students Experiencing Earthquakes
Brief Title: Emotional Freedom Techniques (EFT) on Stress, Anxiety and Depression in University Students Experiencing Earthquakes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7777777
Record Dates: First submitted 2023-12-12; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Emotional Problem; University Students Who Experienced an Earthquake
Keywords: Emotional Freedom Techniques; Earthquake; University Student; Stress; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: EFT will be applied and surveys will be administered to the intervention group. No application will be made to the control group and surveys will be asked.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No application will be performed on the participants in the control group, and as in the intervention group, pre-tests (PSI and STAI) will be carried out immediately after the depression risk determination is made (after the BDI application), and post-tests will be carried out after the interviews are completed. All students in the control group will be reminded of their high scores on the depression scale and will be advised to seek medical help.
- experimental group (Experimental): For applications and information, a computer-assisted zoom program or other online programs that can provide meetings (Google meet, teams program or WhatsApp video call) will be used. The students in the intervention group will be informed about the function and application of EFT, it will be explained practically, and the application steps will be taken. This stage is planned to take approximately 15 minutes.
  Interventions: Other: EFT

INTERVENTIONS:
Other: EFT — EFT
  Arms: experimental group

SUMMARY:
After two earthquakes in Kahramanmaraş Pazarcık in our country, the continuation of long-term aftershocks caused repetition of psychological problems and difficulties in recovery. Social and spiritual support plays a key role in the post-traumatic recovery period. It is necessary to use psychological support methods that can be applied in a short time and whose effect can be observed in a short time in the spiritual healing and healing of traumas. The emotional freedom technique (EFT) is One of the short-term psychotherapeutic techniques and ıt can also be applied online. EFT, which can be easily applied by individuals or professionals after receiving the necessary training; Cognitive therapy, acceptance and commitment therapy combine elements of acupuncture point stimulation, relying on manual stimulation of acupuncture points rather than using acupuncture needles. When we look at the literature, many scientific studies have been found in which the effectiveness of EFT on anxiety, stress and depression has been evaluated, but there has been no randomized controlled study evaluating the effectiveness of EFT online on individuals who have experienced earthquakes. With this project, it is aimed to determine the effect of online Emotional Freedom Techniques (EFT) on stress, anxiety and depression in university students who experienced earthquakes.

This study, which will be carried out as a randomized controlled experimental study, will be carried out between 16.12.2023 and 20.12.2023 by online with university students who score 17 or higher on the Beck Depression Scale. Total of 60 students with depressive symptoms will be recruited to the intervention and control groups, EFT sessions will be applied to the intervention group, and the control group will only be followed. At the beginning of the application, pre-tests (Information Form, Beck Depression Inventory, State Trait Anxiety Inventory, Perceived Stress Inventory) and at the end of the last session, post-tests will be applied for both groups.

With this study, a randomized controlled study will be brought to the literature on the effectiveness of a therapeutic method such as EFT, which is a method that can be used after an earthquake, which is easy to apply, has no cost, and can be accessed online in hard-to-reach areas. Our project will both contribute to the literature and provide short and long-term benefits in practice, in terms of raising awareness of students about important mental problems such as anxiety and depression, which are likely to be experienced after the earthquake, and enabling them to continue their education in a healthy way. It is aimed to present the work planned within the project as a paper in at least one national / international congress. It is aimed to publish in journals within the scope of SCI, SCI-Expanded related to the research area. The results and outputs of the research will be shared in various media (Kırklareli University and Osmaniye Korkut Ata University website and social media accounts).

By determining the stress, anxiety and depression status of university students who have experienced an earthquake, it will be possible to reduce their stress, anxiety and depression with EFT application. The fact that the application used is a short-term, effective and easy psychotherapy method will prevent the disruption of the normal education processes of the students. It will make an economic contribution by reducing the need for psychological drugs that may be needed to reduce the effects of the earthquake.

DETAILED DESCRIPTION:
After two earthquakes in Kahramanmaraş Pazarcık in our country, the continuation of long-term aftershocks caused repetition of psychological problems and difficulties in recovery. Social and spiritual support plays a key role in the post-traumatic recovery period. It is necessary to use psychological support methods that can be applied in a short time and whose effect can be observed in a short time in the spiritual healing and healing of traumas. The emotional freedom technique (EFT) is One of the short-term psychotherapeutic techniques and ıt can also be applied online. EFT, which can be easily applied by individuals or professionals after receiving the necessary training; Cognitive therapy, acceptance and commitment therapy combine elements of acupuncture point stimulation, relying on manual stimulation of acupuncture points rather than using acupuncture needles. When we look at the literature, many scientific studies have been found in which the effectiveness of EFT on anxiety, stress and depression has been evaluated, but there has been no randomized controlled study evaluating the effectiveness of EFT online on individuals who have experienced earthquakes. With this project, it is aimed to determine the effect of online Emotional Freedom Techniques (EFT) on stress, anxiety and depression in university students who experienced earthquakes.

This study, which will be carried out as a randomized controlled experimental study, will be carried out between 16.12.2023 and 20.12.2023 by online with university students who score 17 or higher on the Beck Depression Scale. Total of 60 students with depressive symptoms will be recruited to the intervention and control groups, EFT sessions will be applied to the intervention group, and the control group will only be followed. At the beginning of the application, pre-tests (Information Form, Beck Depression Inventory, State Trait Anxiety Inventory, Perceived Stress Inventory) and at the end of the last session, post-tests will be applied for both groups.

With this study, a randomized controlled study will be brought to the literature on the effectiveness of a therapeutic method such as EFT, which is a method that can be used after an earthquake, which is easy to apply, has no cost, and can be accessed online in hard-to-reach areas. Our project will both contribute to the literature and provide short and long-term benefits in practice, in terms of raising awareness of students about important mental problems such as anxiety and depression, which are likely to be experienced after the earthquake, and enabling them to continue their education in a healthy way. It is aimed to present the work planned within the project as a paper in at least one national / international congress. It is aimed to publish in journals within the scope of SCI, SCI-Expanded related to the research area. The results and outputs of the research will be shared in various media (Kırklareli University and Osmaniye Korkut Ata University website and social media accounts).

By determining the stress, anxiety and depression status of university students who have experienced an earthquake, it will be possible to reduce their stress, anxiety and depression with EFT application. The fact that the application used is a short-term, effective and easy psychotherapy method will prevent the disruption of the normal education processes of the students. It will make an economic contribution by reducing the need for psychological drugs that may be needed to reduce the effects of the earthquake.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older, being a university student, being in the earthquake zone during the earthquake and having experienced the earthquake, not having any infections, wounds or scars in the tapping areas, having a score of 17 or above on the back depression inventory.

Exclusion Criteria:

* Having any problem that prevents communication (such as not knowing Turkish, having impaired hearing, speaking and understanding abilities), being receiving psychiatric treatment (Pharmacotherapy or psychotherapy), not being able to participate online.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
depression | 1 week
  Beck Depression Scale

SECONDARY OUTCOMES:
stress, anxiety | 1 week
  Perceived Stress Scale, State-Trait Anxiety Inventory